CLINICAL TRIAL: NCT01168674
Title: Predictors of Response to Augmentation With Ziprasidone (Geodon®) in Major Depressive Disorder : A 13-week, Double-Blind, Placebo-Controlled, Cross-Over Trial
Brief Title: Predictors of Response to Augmentation With Ziprasidone (Geodon®) in Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Duke University (Other); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 9238
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Depression; Bipolar Disorder
Keywords: Major Depressive Disorder; MDD; Bipolar Disorder; BD; Depression; Major Depressive Disorder with Bipolar features
MeSH Terms: conditions — Depression; Bipolar Disorder; Depressive Disorder, Major | interventions — ziprasidone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Patients are randomized to a sugar pill (placebo), added to their current medications.
  Interventions: Drug: Sugar pill
- Ziprasidone (Active Comparator): Patients are randomized to ziprasidone, added to their current medications.
  Interventions: Drug: ziprasidone

INTERVENTIONS:
Drug: ziprasidone — Ziprasidone will be administered as a pill. The once-daily total daily dose will be 80-160 mg/d of ziprasidone. Dosing will begin at 20 mg BID with an escalation strategy based on target symptoms and tolerability, with a target dose range of 80-160 mg/d. Dose escalations will occur by increments of 20-40 mg weekly.
  Other Names: Geodon
  Arms: Ziprasidone
Drug: Sugar pill — The once-daily total daily dose will be 80-160 mg/d of the sugar pill. Dosing will begin at 20 mg BID with an escalation strategy based on target symptoms and tolerability, with a target dose range of 80-160 mg/d. Dose escalations will occur by increments of 20-40 mg weekly.
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
The primary outcome of this study is to determine if predictors of response can select a population of patients with MDD that is effectively treatable by augmentation with ziprasidone.

Major depressive disorder (MDD) is a broad category, including many forms of depressive illness, including those with only a single major depressive episode, those with episodic recurrence with intervening well states, those with chronic depressive/anxious states without intervening euthymia, and those with manic symptoms that do not meet threshold definitions of full mania/hypomania.

In this heterogenous, large diagnostic definition, important groups of patients do not appear to respond well to antidepressants, and, conversely, based on observational studies, may respond well to neuroleptics. These predictors of response have begun to be identified and may serve to better design studies of neuroleptics in depressive illnesses.

Among these predictors of response in MDD are clinical features that are more similar to bipolar illness than unipolar depression. These include a family history of bipolar disorder, antidepressant-induced mania, highly recurrent depressive episodes (>5), atypical depression, early age of onset of depression (< age 20), failure to respond to antidepressants, and antidepressant tolerance (initial response followed by later loss of response).

The investigators propose to use these predictors to pick out patients that are more likely to respond to Geodon for MDD. This will be the first RCT of these predictors of depressive response applied to neuroleptics.

DETAILED DESCRIPTION:
This will be a three-site, block randomized (1:1 ratio) double-blind, placebo-controlled prospective cross-over study with 50 subjects. Patients will be randomized to receiving ziprasidone-washout-placebo or placebo- washout-ziprasidone for 13-weeks.

Primary and Secondary and safety outcomes: The primary outcome measure will be change from baseline Montgomery-Asberg Depression Rating Scale (MADRS) score to end of treatment. Safety outcomes will be determined by spontaneously reported adverse events on the case report form.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years.
2. If female, nonpregnant/nonlactating
3. If a sexually active female of reproductive potential, must be using adequate contraception (i.e., oral contraceptives, barrier protection, or prior tubal ligation)
4. Currently meets DSM-IV criteria for a major depressive episode, non-psychotic.
5. Having at least 3 of the following criteria listed for predictors of depressive response to neuroleptics: a family history of bipolar disorder, antidepressant-induced mania, highly recurrent depressive episodes (>5), atypical depression, early age of onset of depression (< age 20), failure to respond to antidepressants, and antidepressant tolerance (initial response followed by later loss of response). Inadequate response to antidepressants is identified as follows: having a score of ≥14 on the 17-item HAMD or a CGI-S score of ≥ 3 after a retrospective confirmation of an adequate trial of a single antidepressant (defined as a ≥ 6-week trial of acceptable therapeutic dose [≥ 40 mg of fluoxetine, paroxetine or citalopram, 20 mg of escitalopram, 60 mg of duloxetine, 37.5 mg of paroxetine CR, 150 mg of sertraline, 100 mg of fluvoxamine, 225 mg of venlafaxine XR, 30 mg of mirtazapine, 300 mg of bupropion, 75 mg of nortriptyline, 20 mg of protriptyline, 100 mg of amitriptyline or imipramine)

Exclusion Criteria:

1. Bipolar depression
2. Sensitivity to or failure to respond to ziprasidone by history or ziprasidone use in previous 3 months
3. Active substance abuse or dependence in the previous 3 month
4. Psychotic disorders
5. Serious suicidality as evidenced by score of 3 or greater on suicide item of MADRS
6. Medically unstable as judged by study investigators
7. Lack of capacity to provide informed, written, consent to investigators
8. Previous diagnosed cardiac arrhythmias

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Ghaemi, MD MPH, Principal Investigator — Tufts Medical Center; Ashwin Patkar, MD, Principal Investigator — Duke; Meera Narasimhan, MD, Principal Investigator — University of South Carolina; Prakash Masand, MD, Principal Investigator — Duke

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-washout-ziprasidone: Placebo : The once-daily total daily dose will be 80-160 mg/d of the sugar pill. Dosing will begin at 20 mg BID with an escalation strategy based on target symptoms and tolerability, with a target dose range of 80-160 mg/d. Dose escalations will occur by increments of 20-40 mg weekly. This will be 6 weeks and then followed by a one week washout and then cross over to the other arm, Ziprazidone, for another 6 weeks, using same dosing techniques.
- Ziprasidone-washout-placebo: ziprasidone : Ziprasidone will be administered as a pill. The once-daily total daily dose will be 80-160 mg/d of ziprasidone. Dosing will begin at 20 mg BID with an escalation strategy based on target symptoms and tolerability, with a target dose range of 80-160 mg/d. Dose escalations will occur by increments of 20-40 mg weekly. This will be 6 weeks and then followed by a one week washout and then cross over to the other arm, Placebo, for another 6 weeks, using same dosing techniques.
Period: Overall Study
Arm/Group | Placebo-washout-ziprasidone | Ziprasidone-washout-placebo
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to either placebo followed by ziprasidone crossover, or ziprsidone followed by placebo crossover.
Arm/Group | All Study Participants
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: MADRS Improvement Over 6 Weeks
Description: Montgomery Asberg Depression scale improvement was assessed in two 6 week crossover periods.
  Minimum score on MADRS is 0, the maximum is 60. Higher scores represent a worse outcome, i.e., greater severity of depressive symptoms.
  Scores of about 20 and above are generally seen as consistent with being in a full major depressive episode.
  No subscales were used or combined.
Time Frame: 13 weeks (Two 6 week periods plus a one week washout)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Subjects randomized to placebo in either the initial or crossover phase
- Ziprasidone: Subjects randomized to ziprasidone in either the initial or crossover phase.
Arm/Group | Placebo | Ziprasidone
Number analyzed (Participants) | 49 | 49
units on a scale | 10.0 (10.3) | 6.7 (8.2)
Statistical Analysis 1: Comparison: Placebo vs Ziprasidone; Linear mixed effects regression model; Test type: Superiority or Other; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = 1.57, Standard Deviation 1.67 — The report is of the mean MADRS difference between ziprasidone versus placebo after linear mixed regression, correcting for confounding effects of order of treatment as well as other identified potential confounders

2. Secondary Outcome: Predictors of Bipolarity to Define the Study Population
Description: The specific bipolarity predictors in patients with MDD were assessed.
Time Frame: 13 weeks
Population: The most common predictor was antidepressant tolerance, as reported below in 37 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | All Study Participants
Number analyzed (Participants) | 49
percentage of subjects
  Antidepressant tolerance | 75.0
  Antidepressant nonresponse | 73.5
  Highly recurrent depressive episodes | 72.3
  Atypical depression | 52.9
  Family history of bipolar disorder | 46.0
  Early age of onset | 47.6
  Antidepressant-induced mania | 8.8

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: Adverse events are reported as ziprasidone arm events over placebo given the crossover nature of the study.
Groups:
- Placebo: Placebo administered double-blind.
- Ziprasidone: Active ziprasidone administered double-blind.
Arm/Group | Placebo | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/49
Other Adverse Events (participants affected / at risk) | 0/49 | 21/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Ziprasidone (N=49)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Ziprasidone (N=49)
sedation (Nervous system disorders) | 0 (0) | 8 (8)
nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
dry mouth (Nervous system disorders) | 0 (0) | 4 (4)
constipation (Gastrointestinal disorders) | 0 (0) | 5 (5)

LIMITATIONS AND CAVEATS:
All crossover studies have the limitation of order effects: the order in which treatments were given could impact the results. The definition of bipolarity predictors also may not have effectively identified groups correctly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No